CLINICAL TRIAL: NCT05843968
Title: Rituximab Versus Mycophenolate Mofetil in Children With Steriod-dependent Nephrotic Syndrome: A Single-center, Randomized Controlled Trial
Brief Title: Efficacy and Safety of Rituximab Versus Mycophenolate Mofetil in Children With Steroid-dependent Nephrotic Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Haiping Yang, Associate Director of Nephrology, Children's Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYang
Record Dates: First submitted 2023-04-08; First posted 2023-05-06 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Nephrotic Syndrome in Children
Keywords: Nephrotic Syndrome; Rituximab; Mycophenolate Mofetil
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Rituximab; Mycophenolic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rituximab (Experimental): 2 doses of rituximab 375 mg/m^2 (Maximum 500mg/day)at 6 months intervals
  Interventions: Drug: Rituximab
- Mycophenolate Mofetil (Active Comparator): MMF 20~30mg/kg/day，BID
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Rituximab — 2 doses of rituximab 375 mg/m^2(maximum 500mg/day) at 6 months intervals.
  Half an hour before rituximab infusion: oral acetaminophen 15mg/kg, oral or intramuscular antihistamine, methylprednisolone 2mg/kg IV. Trimethoprim-sulfamethoxazole should be administered orally from the initiation of rituximab therapy until peripheral-blood B cell recovery to prevent pneumocystis infection.
  Other Names: Rituximab Injection
  Arms: Rituximab
Drug: Mycophenolate Mofetil — Mycophenolate Mofetil 20-30 mg/kg/day BID,then adjust the dosage of drugs(maximum 2g/day) to maintian the concentration for MPA-AUC is 30-50μg.h/ml. Total duration:1year.
  Steroids dose:1.5mg/kg(maximum 40mg) qod for 2 weeks and gradually taper by 0.3 mg/kg every 2 weeks
  Other Names: Mycophenolate Mofetil Dispersible tablets
  Arms: Mycophenolate Mofetil

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of rituximab(RTX) and mycophenolate mofetile(MMF) in the treatment of children with low-dose steroid-dependent nephrotic syndrome(SDNS).

DETAILED DESCRIPTION:
Idiopathic nephrotic syndrome（INS） is the most common glomerular disease in childhood. Currently, steroids are the primary treatment, but there are significant steroid-related toxicity, such as growth disorders, behavior changes, obesity, Cushing's syndrome, eye disease, osteoporosis, etc.

Both MMF and RTX have been shown to be effective in the treatment of SDNS, and there is a lack of prospective controlled studies to explore the optimal treatment regimen for low-dose SDNS. Therefore, the investigators will conduct a single-center, randomized controlled trial to evaluate the efficacy and safety of twice-daily rituximab(RTX) versus mycophenolate mofetil(MMF) in the treatment of children with low-dose steroid-dependent nephrotic syndrome(SDNS).

After the start of the study, all participants will be screened consecutively and eligible participants will be included in the study. Bias of potential influencing factors will be addressed by inclusion as covariates in the statistical analysis. Independent clinical site monitoring to ensure the safety and integrity of clinical data while patients adhere to the study protocol will focus on source data documentation, strict adherence to data correctness and study procedures, such as randomization and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children with a definite diagnosis of SDNS are included in the study during relapse treatment.
* Age 3-16 years.
* Steroid dependent dose≤0.3mg/kg/day.
* Cumulative steroid use for ≥6 months.
* Ability to swallow tablet.
* Guardians understand the characteristics and personal consequences of clinical trial.
* Guardians willing to give informed written consent.

Exclusion Criteria:

* Diagnosis of secondary NS, such as secondary to lupus nephritis, hepatitis B-related nephritis, purpura nephritis, etc.
* Anti-neutrophil cytoplasmic antibodies(ANCA) positive or complement C3 level decreased.
* Diagnosis of hereditary nephrotic syndrome.
* Full dose of prednisone (2mg/kg/day, maximum 60mg) are used for 14 days after relapse and urine protein don't turn negative.
* Estimated glomerular filtration rate (eGFR) <90mL/min per 1.73m^2 at study entry.
* Those who with a known allergy to Mycophenolate Mofetil and their excipients or to Rituximab and its excipients.
* Those who refuse to participate in the trial.
* Those who participate other clinical trials.
* Those who with positive HBV serological markers (HBsAg or/and HBeAg or/and HBcAb), HCV positive patients or patients with abnormal liver function (ALT,AST,or bilirubin>2 or more times the upper limit of the normal range and persistently elevated for 2 weeks).
* Severe leukopenia (white blood cells<3.0×10^9), severe anemia (hemoglobin<90g/l), and thrombocytopenia (platelets<100×10^9) at study entry.
* History of pancreatitis or definite gastrointestinal ulcers and/or gastrointestinal bleeding within 6 months.
* Those who with congenital or acquired immune deficiency, or with active tuberculosis, active CMV and other infections.
* Those who with other serious physical or mental illnesses.
* History of malignant tumor within 5 years.
* Those who with congenital heart disease, arrhythmia, heart failure and other serious cardiovascular diseases.
* Those who with serious infections requiring intravenous antibiotics.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Estimated)
Dates: Start 2023-01-29 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
12-month relapse-free survival rate | 12 months
  The rate of no relapse within 12 months.

SECONDARY OUTCOMES:
6-month relapse-free survival | 6 months
  Relapse-free survival within 6 months.
6-month relapse-free survival rate | 6 months
  The rate of no relapse within 6 months.
12-month relapse-free survival | 12 months
  Relapse-free survival within 12 months.
Proportion of frequent relapses | Months 6,12
  The proportion of frequent relapses.Frequent relapsing NS:≥2 relapses per 6 months within 6 months of disease onset or ≥4 relapses per 12 months in any subsequent 12-month period.
Cumulative steroid dosage | 12 months
  The total dosage of steroid from the beginning to the end of the trial.
Number of relapses within 0-12,0-6, and 7-12 months | 12 months
  Number of relapses within 0-6 months,7-12 months, and total within 0-12 months.
Time of first relapse | 12 months
  The first time to relapse after patients taking part in this study.
Adverse event | 12 months
  It is a binary variable(1/0).The varibale would be setted as "1" if any adverse events occours including obesity, hypertrichosis, psychological disorders,glaucoma,neutropenia,hypogammaglobulinemia, rituximab-related lung injury, fatal hepatitis reactivation, multifocal leukoencephalopathy,severe diarrhea, severe infection. Adverse events graded according to Common Terminology Criteria For Adverse Events (CTCAE v4.0）
Proportion of participants who discontinued steroids | 12 months
  Proportion of participants who discontinued steroids at 12 months
Height standard deviation score(SDS) | months 0,6,12
  SDS of height at 6 and 12 months, absolute and relative changes in SDS from baseline to 12 months.
Body mass index(BMI) | Months 0,6,12
  Weight and height will be combined to report BMI in kg/m^2. BMI at 6 and 12 months, absolute and relative changes in BMI from baseline to 12 months.
Quality of life score | Baseline to 12 months
  The researchers assess the quality of life of the participants useing Pediatric Quality of Life Inventory (PedsQL).
Cost of treatment | 12 months
  The researchers calculate their cost during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Larkins NG, Hahn D, Liu ID, Willis NS, Craig JC, Hodson EM. Non-corticosteroid immunosuppressive medications for steroid-sensitive nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Nov 8;11(11):CD002290. doi: 10.1002/14651858.CD002290.pub6. PMID 39513526